CLINICAL TRIAL: NCT02028806
Title: Phase Ⅱ Trial to Investigate the Efficacy and Safety of mFOLFIRINOX in Patients With Metastatic Pancreatic Cancer in China
Brief Title: mFOLFIRINOX as First-Line Chemotherapy in Treating Chinese Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yuhong Li (Other)
Responsible Party: Sponsor-Investigator, Yuhong Li, MD, Ph D, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAN-321
Record Dates: First submitted 2014-01-01; First posted 2014-01-07 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Oxaliplatin; Irinotecan; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFIRINOX (Experimental): Patients will receive mFOLFIRINOX every 2 weeks: Oxaliplatin 65 mg/m2 IV over 3 hours on Day 1; Irinotecan 150 mg/m2 IV over 90 minutes on Day 1; Leucovorin(l-LV) 200 mg/m2 IV over 2 hours on Day 1; followed by 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion.
  Interventions: Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: mFOLFIRINOX — Patients will receive mFOLFIRINOX every 2 weeks: Oxaliplatin 65 mg/m2 IV over 3 hours on Day 1; Irinotecan 150 mg/m2 IV over 90 minutes on Day 1; Leucovorin(l-LV) 200 mg/m2 IV over 2 hours on Day 1; followed by 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion.
  Other Names: Oxaliplatin; Irinotecan; Leucovorin; 5-Fluorouracial

SUMMARY:
This phase Ⅱ study was designed to evaluate the efficacy and safety of mFOLFIRINOX as first-line treatment for metastatic pancreatic cancer in China.

DETAILED DESCRIPTION:
Although FOLFIRINOX regimen was recently presented to be effective for metastatic pancreatic cancer in selected patients who have good physical condition, there is still insufficient evidence on this regimen in treating patients with metastatic pancreatic cancer in China. Since for many tumors, different races may show different responses to the same regimen, we design this open, multicenter phase Ⅱ study to evaluate the the efficacy and safety of mFOLFIRINOX as first-line treatment for metastatic pancreatic cancer in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients have provided a signed Informed Consent Form
* ECOG performance status of 0-1
* BMI ≥ 18.5
* Age: 18-65 years old
* Histologically confirmed diagnosis of metastatic pancreatic cancer
* No prior palliative chemotherapy
* Measurable disease in at least 1 diameter by CT scan or MRI as per RECIST 1.1 criteria
* Life expectancy ≥ 3 months
* Patient has adequate bone marrow and organ function

  * Absolute Neutrophil Count (ANC) ≥ 2.0 x 109/L
  * Platelets ≥ 90 x 109/L
  * Hemoglobin ≥ 90 g/L
* Patient has adequate liver function

  * AST and ALT not more than 2.5 times ULN (not more than 5.0 times ULN if there is liver metastasis)
  * Serum bilirubin ≤ 1.2 x ULN
* Creatinine ≤ 1.25 times ULN
* Good compliance

Exclusion Criteria:

* Pregnant or lactating women
* Brain metastasis or only with bone metastasis.
* Patients with severe gastrointestinal hemorrhage which need frequent blood transfusions.
* Refuse to take appropriate contraceptive measures (including male patients).
* Allergic to Oxaliplatin, Irinotecan, Leucovorin or 5-Fluorouracil.
* Severe systemic disease out of control such as unstable or uncompensated respiratory, cardiac, liver, renal diseases.
* Patient has a concurrent malignancy or has a malignancy within 5 years of study enrollment, (with the exception of non-melanoma skin cancer or cervical carcinoma in situ).
* Psychiatric illness that would prevent the patient from giving informed consent.
* Patient is concurrently using other antineoplastic agent
* Patient has used investigational antineoplastic agent within 4 weeks prior to entry.
* Known HIV-positivity.
* No history of chronic diarrhea, nausea or vomit.
* No ≥ grade 2 sensory peripheral neuropathy.
* A history of transmural myocardial infarction (within 6 months prior to entry), congestive heart failure, and unstable angina.
* Infectious disease or inflammation with body temperature ≥ 38 ℃.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Disease control rate | Up to 24 weeks

SECONDARY OUTCOMES:
Progression free survival | From the date of first drug administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
Overall survival | From the date of first drug administration until the date of death, assessed up to 60 months
Number of participants with AEs and SAEs as a measure of Safety | Each follow up visit, assessed up to 24 weeks
  Safety data will be assessed at each study visit using NCI CTCAE version 3.0
EORTC QLQ-C30 | Each follow up visit, assessed up to 24 weeks
  Quality of life will be assessed at each study using EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Overall Officials: Li Yuhong, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wang ZQ, Zhang F, Deng T, Zhang L, Feng F, Wang FH, Wang W, Wang DS, Luo HY, Xu RH, Ba Y, Li YH. The efficacy and safety of modified FOLFIRINOX as first-line chemotherapy for Chinese patients with metastatic pancreatic cancer. Cancer Commun (Lond). 2019 May 8;39(1):26. doi: 10.1186/s40880-019-0367-7. PMID 31068222